CLINICAL TRIAL: NCT01479140
Title: Prospective Registry of Young Women With MI: Evaluating the Prevalence and Long-term Impact of Non-atherosclerotic CAD (PRYME)
Brief Title: Prevalence and Long-term Impact of Non-atherosclerotic CAD
Acronym: PRYME
Status: Completed | Type: Observational
Sponsor: Cardiology Research UBC (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jacqueline Saw, MD, Principal Investigator, Dr. Jackie Saw, Vancouver General Hospital
Other Study IDs: H11-03186
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; dissection; coronary Fibromuscular Dysplasia; coronary ectasia; atherosclerotic Coronary Artery Disease; coronary vasculitis; coronary embolism; congenital coronary anomaly
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite a relatively high prevalence of non-atherosclerotic coronary artery disease (NACAD) among young women, the majority of these abnormalities were misdiagnosed in this population, and thus treatments were not targeted adequately in this patient population. Furthermore, the short and long-term cardiovascular outcomes of young women with NACAD have not been evaluated. Given the importance of NACAD in young women, the challenges of diagnosis and subsequent treatment, and unknown outcomes with NACAD, we propose a prospective registry to further evaluate this population. We propose to evaluate young women (age < or equal to 55) presenting with myocardial infarction (MI) prospectively, to diagnose the etiology of MI differentiating atherosclerotic versus NACAD, to correlate the prevalence of FMD in other vascular territory, and to evaluate the long-term outcome of young women with NACAD in comparison to those with atherosclerotic CAD over a 5-year follow-up.

DETAILED DESCRIPTION:
All women aged 55 or younger having a coronary angiogram for acute coronary syndrome (ACS) will be approached prior to their procedure. A pregnancy test will be performed (standard for pre-menopausal women due to potential radiation exposure). If the cause of the heart attack is uncertain (eg no obvious infarct-related narrowing or occlusion), intravascular ultrasound or optimal coherence tomography will be performed within the context of the angiogram to better view the artery wall. A picture of the iliac and renal arteries will be accomplished by aortography (one dye shot down the aorta); in the case that the renal arteries are not well visualized, selective renal angiography will be performed (catheter at the entry to the renal artery). In the case of suspected non-atherosclerotic abnormalities, a head CT angiogram wil be performed. Referral to appropriate specialists for detected abnormality will occur. If symptoms continue, the subject will be followed by a cardiologist. A research coordinator will contact the subject at 1, 6 and 12 months and then annually to collect data on medications, hospitalization and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 55 or younger with a troponin positive acute coronary syndrome (ST and non-ST elevation myocardial infarction or Acute Coronary Syndrome (ACS)) having a coronary angiogram
* negative pregnancy test for women of child bearing age

Exclusion Criteria:

* Creatinine clearance <50
* not willing to undergo an angiogram
* troponin negative ACS

Ages: 19 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 55 or younger with a troponin positive acute coronary syndrome (ST and non-ST elevation myocardial infarction or Acute Coronary Syndrome (ACS)) having a coronary angiogram
  Negative pregnancy test
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-12; Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Evaluate the etiology of MI | 5 years
  To evaluate the etiology of myocardial infarction among young women (age < or equal to 55) based on angiographic and adjunctive imaging by core laboratory assessment
Evaluate the relative distribution of normal coronary arteries, atherosclerotic, and non-atherosclerotic CAD in this population of young women with MI | 5 years
  Evaluate the relative distribution of normal coronary arteries, atherosclerotic, and non-atherosclerotic CAD in this population of young women with MI
to screen for the prevalence of SCAD and coronary FMD as the predominant non-atherosclerotic cause for MI in young women | 5 years
  to screen for the prevalence of SCAD and coronary FMD as the predominant non-atherosclerotic cause for MI in young women

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Saw, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada